CLINICAL TRIAL: NCT03418493
Title: A Phase 1 Randomized, Placebo-Controlled Study of LY3316531 in Healthy Subjects and an Open-Label, Single-Dose Study in Patients With Psoriasis
Brief Title: A Study of LY3316531 in Healthy Participants and in Participants With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16666; I9H-MC-FFAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3316531 (Part A) (Experimental): Participants received single doses of 3 milligrams (mg), 15 mg, 75 mg, 300 mg, 900 mg, or 2000 mg LY3316531 administered Intravenously (IV), or 300 mg LY3316531 administered Subcutaneously (SC).
  Interventions: Drug: LY3316531 - IV; Drug: LY3316531 - SC
- Placebo (Part A) (Placebo Comparator): Placebo matching LY3316531 administered IV.
  Interventions: Drug: Placebo - IV
- LY3316531 (Part B) (Experimental): Participants received 3 doses of 2000 mg LY3316531 administered IV (1 dose every 4 weeks).
  Interventions: Drug: LY3316531 - IV
- Placebo (Part B) (Placebo Comparator): Placebo matching LY3316531 administered IV.
  Interventions: Drug: Placebo - IV
- LY3316531 (Part C) (Experimental): Participants with psoriasis received single doses of 300 mg LY3316531 administered IV.
  Interventions: Drug: LY3316531 - IV

INTERVENTIONS:
Drug: LY3316531 - IV — Administered IV.
  Arms: LY3316531 (Part A); LY3316531 (Part B); LY3316531 (Part C)
Drug: LY3316531 - SC — Administered SC.
  Arms: LY3316531 (Part A)
Drug: Placebo - IV — Administered IV.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate how well LY3316531 is tolerated and what side effects may occur in healthy participants and participants with psoriasis. The study drug will be administered either subcutaneously (SC) (under the skin) or intravenously (IV) (into a vein in the arm).

This is a three-part study. Participants will enroll in only one part. Parts A and B are for healthy participants and Part C is for participants with psoriasis. Participation could last between 16 and 57 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants

  * Are overtly healthy males or females, as determined by medical history and physical examination
  * Females must be of non-childbearing potential
  * Are between 18 and 64 years of age, inclusive, at screening
  * Have a body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m²) inclusive
  * Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Psoriasis Participants:

  * Chronic plaque psoriasis based on an investigator confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to baseline
  * Meet psoriasis disease activity criteria
  * Are at least 18 years of age
  * Have a minimum body weight of 50 kilograms (kg)

Exclusion Criteria:

* Healthy and Psoriasis Participants

  * Have known or ongoing neuropsychiatric disorders
  * Have received live vaccine(s) (included attenuated live vaccines) within 28 days of screening or intend to during the study
  * Have had any malignancy within the past 5 years except for basal cell or squamous cell epithelial carcinomas of the skin that have been resected with no subsequent evidence of recurrence for at least 3 years prior to screening and cervical carcinoma in situ with no evidence of recurrence within 5 years prior to baseline
  * Show evidence of active or latent tuberculosis (TB)
  * Have presence of significant uncontrolled cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic or neuropsychiatric disorders or abnormal laboratory values at screening that, in the opinion of the investigator, pose an unacceptable risk to the participant if participating in the study or of interfering with the interpretation of data
* Psoriasis Participants Only:

  * Have received treatment with biologic therapies for psoriasis (such as monoclonal antibodies, including marketed or investigational biologic therapy)
  * Prior or current use of biologics for indications other than psoriasis may be allowed with sponsor approval
  * Have received systemic nonbiologic psoriasis therapy within 28 days of baseline
  * Have received topical psoriasis treatment within 14 days of baseline

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3316531 in Healthy Participants and in Participants With Psoriasis — https://www.lillytrialguide.com/en-US/studies/psoriasis/FFAA#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consists of three parts:
  * Part A (Single-Ascending Dose (SAD) in healthy participants)
  * Part B (Multiple-dose in healthy participants) and
  * Part C (Single dose in psoriasis participants)
Groups:
- Placebo - Part A: Participants received single IV doses of Placebo.
- 3 mg LY3316531 IV - Part A: Participants received single doses of 3 milligrams (mg) LY3316531 administered Intravenously (IV).
- 15 mg LY3316531 IV - Part A: Participants received single doses of 15 mg LY3316531 administered IV.
- 75 mg LY3316531 IV - Part A: Participants received single doses of 75 mg LY3316531 administered IV.
- 300 mg LY3316531 IV - Part A: Participants received single doses of 300 mg LY3316531 administered IV.
- 300 mg LY3316531 SC- Part A: Participants received single doses of 300 mg LY3316531 administered Subcutaneously (SC).
- 900 mg LY3316531 IV - Part A: Participants received single doses of 900 mg LY3316531 administered IV.
- 2000 mg LY3316531 IV - Part A: Participants received single doses of 2000 mg LY3316531 administered IV.
- Placebo - Part B: Participants received 3 doses of Placebo administered IV (1 dose every 4 weeks).
- 2000 mg LY3316531 IV - Part B: Participants received 3 doses of 2000 mg LY3316531 administered IV (1 dose every 4 weeks).
- 300 mg LY3316531 IV - Part C: Participants with psoriasis received single doses of 300 mg LY3316531 administered IV.
Period: Overall Study
Arm/Group | Placebo - Part A | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A | Placebo - Part B | 2000 mg LY3316531 IV - Part B | 300 mg LY3316531 IV - Part C
Started | 11 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 8
Completed | 10 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 5 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Part A | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A | Placebo - Part B | 2000 mg LY3316531 IV - Part B | 300 mg LY3316531 IV - Part C | Total
Number analyzed (Participants) | 11 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 8 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 8 | 63
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 1 | 3 | 17
  Male | 7 | 2 | 2 | 4 | 5 | 6 | 4 | 5 | 1 | 5 | 5 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 2 | 4 | 2 | 2 | 2 | 1 | 0 | 0 | 17
  Not Hispanic or Latino | 9 | 2 | 2 | 4 | 2 | 4 | 4 | 4 | 1 | 6 | 8 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 5 | 2 | 0 | 3 | 1 | 0 | 2 | 2 | 0 | 2 | 4 | 21
  White | 5 | 1 | 2 | 3 | 5 | 4 | 3 | 4 | 2 | 2 | 3 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 8 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality is reported in the Reported Adverse Events module.
  An SAE is any adverse event from this study that results in 1 of the following:
  1. Death
  2. Initial or prolonged inpatient hospitalization
  3. A life-threatening experience (that is, immediate risk of dying)
  4. Persistent or significant disability/incapacity
  5. Congenital anomaly/birth defect
  6. Important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above.
Time Frame: Pre-dose up to 1 year after administration of study drug
Population: All randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Part A | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A | Placebo - Part B | 2000 mg LY3316531 IV - Part B | 300 mg LY3316531 IV - Part C
Number analyzed (Participants) | 11 | 3 | 3 | 6 | 6 | 6 | 6 | 6 | 2 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Secondary Outcome: Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3316531
Description: PK: Cmax of LY3316531. Under time frame, hours was abbreviated as "hrs."
Time Frame: Pre-dose, Days 1 (End of infusion [IV], 2 hrs after start of infusion [IV], 6 hrs after start of infusion [IV] or injection [SC]), 2 (24 hrs after start of infusion [IV] or injection [SC]), 4, 8, 11 (SC only), 15, 22, 29, 43, 57, 71, 85 post- dose
Population: All randomized participants in Part A who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6
micrograms per milliliter (μg/mL) | 1.27 (18) | 9.94 (26) | 32.7 (22) | 115 (11) | 27.2 (30) | 453 (14) | 808 (15)

3. Secondary Outcome: Part B: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3316531
Description: PK: Cmax of LY3316531 following the Day 57 dose.
Time Frame: Days 57 (Pre-dose, end of infusion), 58, 60, 64, 67, 71, 78, and 85
Population: All randomized participants in Part B who received study drug on Day 57 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 2000 mg LY3316531 IV - Part B
Number analyzed (Participants) | 5
μg/mL | 876 (14)

4. Secondary Outcome: Part C: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3316531
Description: PK: Cmax of LY3316531.
Time Frame: Pre-dose, Days 1 (End of infusion, 2 hrs after start of infusion, 6 hrs after start of infusion), 2 (24 hrs after start of infusion), 4, 8, 15, 22, 29, 43, 57, 71, 85, and 113 post-dose
Population: All randomized participants in Part C who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 300 mg LY3316531 IV - Part C
Number analyzed (Participants) | 8
μg/mL | 124 (19)

5. Secondary Outcome: Part A: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3316531 From Time Zero to Infinity - AUC(0-∞)
Description: Area Under the Concentration Versus Time Curve (AUC) of LY3316531 From Time Zero to Infinity - AUC(0-∞).
Time Frame: as for outcome 2
Population: All randomized participants in Part A who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours per milliliter(μg*h/mL)
Arm/Group | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 6
micrograms*hours per milliliter(μg*h/mL) | 401 (7) | 3050 (23) | 12,700 (19) | 46,900 (10) | 25,800 (27) | 181,000 (25) | 319,000 (31)

6. Secondary Outcome: Part B: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3316531 Over the Dosing Interval (Tau) - AUCtau
Description: AUC of LY3316531 over the dosing interval (tau = 672 h = 28 days) following the Day 57 dose.
Time Frame: Days 57 (Pre-dose, end of infusion), 58, 60, 64, 67, 71, 78, and 85
Population: All randomized participants in Part B who received study drug on Day 57 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 2000 mg LY3316531 IV - Part B
Number analyzed (Participants) | 5
μg*h/mL | 258,000 (2)

7. Secondary Outcome: Part C: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3316531 From Time Zero to Infinity - AUC(0-∞)
Description: Area Under the Concentration Versus Time Curve (AUC) of LY3316531 From Time Zero to Infinity - AUC(0-∞).
Time Frame: as for outcome 4
Population: All randomized participants in Part C who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 300 mg LY3316531 IV - Part C
Number analyzed (Participants) | 8
μg*h/mL | 39,500 (28)

ADVERSE EVENTS:
Time Frame: Up To 1 Year
Description: All randomized participants who received study drug.
Arm/Group | Placebo - Part A | 3 mg LY3316531 IV - Part A | 15 mg LY3316531 IV - Part A | 75 mg LY3316531 IV - Part A | 300 mg LY3316531 IV - Part A | 300 mg LY3316531 SC- Part A | 900 mg LY3316531 IV - Part A | 2000 mg LY3316531 IV - Part A | Placebo - Part B | 2000 mg LY3316531 IV - Part B | 300 mg LY3316531 IV - Part C
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 1/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/11 | 1/3 | 1/3 | 1/6 | 1/6 | 5/6 | 2/6 | 1/6 | 1/2 | 4/6 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Part A (N=11) | 3 mg LY3316531 IV - Part A (N=3) | 15 mg LY3316531 IV - Part A (N=3) | 75 mg LY3316531 IV - Part A (N=6) | 300 mg LY3316531 IV - Part A (N=6) | 300 mg LY3316531 SC- Part A (N=6) | 900 mg LY3316531 IV - Part A (N=6) | 2000 mg LY3316531 IV - Part A (N=6) | Placebo - Part B (N=2) | 2000 mg LY3316531 IV - Part B (N=6) | 300 mg LY3316531 IV - Part C (N=8)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Part A (N=11) | 3 mg LY3316531 IV - Part A (N=3) | 15 mg LY3316531 IV - Part A (N=3) | 75 mg LY3316531 IV - Part A (N=6) | 300 mg LY3316531 IV - Part A (N=6) | 300 mg LY3316531 SC- Part A (N=6) | 900 mg LY3316531 IV - Part A (N=6) | 2000 mg LY3316531 IV - Part A (N=6) | Placebo - Part B (N=2) | 2000 mg LY3316531 IV - Part B (N=6) | 300 mg LY3316531 IV - Part C (N=8)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maternal exposure before pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT03418493/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT03418493/SAP_001.pdf